CLINICAL TRIAL: NCT05955131
Title: Formulación de Productos de panificación Suplementados Con Harina de Porotos Nativos Chilenos Para Disminuir Respuestas glicémicas Postprandiales y agregación Plaquetaria en Personas Mayores: Un Estudio Piloto
Brief Title: Bread Supplemented With Chilean Beans to Decrease Postprandial Glycoxidative Responses: A Pilot Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Talca (Other)
Collaborators: Interuniversity Center for Healthy Aging (Unknown); Centro de Estudios en Alimentos Procesados (Other); Clínica Fleming de Talca (Unknown)
Responsible Party: Principal Investigator, Felipe Ávila Concha, Asociate Professor, University of Talca
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CIES 002
Record Dates: First submitted 2023-06-27; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Aging
Keywords: Oxidative stress; Glycoxidation; Advanced glycation end products; Aging; Bread; Antioxidants; Fiber; Platelet aggregation

STUDY DESIGN:
Intervention Model Description: This study involves an acute nutritional intervention with crossover design, in which each volunteer will eat one out of tree meals (control bread, supplemented bread or glucose), randomly, once by week. Blood samples will be taken at 0min and 30, 60 and 120 min postprandial. The volunteers will complete their participation after the intake of the three meals, hence, their participation in the study will finish after 3 weeks.
Who Masked: Investigator
Masking Description: Blood samples will be codified, and the keys will be saved by Felipe Ávila. The personal in charge of the blood analyses (quantification of methylglyoxal and 3-deoxyglucosone) will register their results using the codes and therefore will not know the type of sample analyzing or the volunteer that provided the sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Bread (Other): Subjects will eat control bread, in an amount containing 50g of carbohydrates
  Interventions: Other: Nutritional acute postprandial intervention: Control bread
- Bread Supplemented with Chilean Beans (Experimental): Subjects will eat bread supplemented with Chilean native beans at 30% w/w, in an amount containing 50g of carbohydrates
  Interventions: Other: Nutritional acute postprandial intervention: bread suppelmented with Chilean beans
- Glucose control (Other): Subjects will drink glucose, in an amount containing 50g of carbohydrates
  Interventions: Other: Nutritional acute postprandial intervention: Control glucose

INTERVENTIONS:
Other: Nutritional acute postprandial intervention: Control bread — Volunteers will arrive at fasting and blood samples (aprox. 5mL) will be obtained before (0 min) and after the intake (10 min of intake) an amount of control bread containing 50g of carbohydrates, venous blood samples for determination of insulin, methyglyoxal, 3-deoxyglucosone and platelet aggregation will be collected at 30, 60, 90 and 120 mn postprandial. In addition, capillary slood will be obtained at 0, 15, 30, 60, 90 and 120 postprandial for glycemia determination
  Arms: Control Bread
Other: Nutritional acute postprandial intervention: bread suppelmented with Chilean beans — Volunteers will arrive at fasting and blood samples (aprox. 5mL) will be obtained before (0 min) and after the intake (10 min of intake) an amount of supplemented bread containing 50g of carbohydrates, venous blood samples for determination of insulin, methyglyoxal, 3-deoxyglucosone and platelet aggregation will be collected at 30, 60, 90 and 120 mn postprandial. In addition, capillary slood will be obtained at 0, 15, 30, 60, 90 and 120 postprandial for glycemia determination.
  Arms: Bread Supplemented with Chilean Beans
Other: Nutritional acute postprandial intervention: Control glucose — Volunteers will arrive at fasting and capillary blood samples will be obtained before (0 min) and after the intake an amount of control glucose containing 50g of this monosscharide (10 min of intake), capillary slood will be also obtained at 15, 30, 60, 90 and 120 postprandial for glycemia determination.
  Arms: Glucose control

SUMMARY:
The goal of this trial is to assess in healthy subjects between 60 and 70 years the effect of glycemic and glycoxidative postprandial responses and platelet aggregation after intake of bread supplemented with Chilean beans flour when compared with a non supplemented control. The main questions to answer are:

* It is possible to decrease postprandial glycemic and glycoxidative responses by means of the intake of bread supplemented with Chilean beans flour when compared to the intake of a control bread non supplemented in healthy elderly persons?
* How is affected the platelet aggregation process during postprandial state after intake of bread supplemented with Chilean beans flour, when compared to the intake of a control bread non supplemented in healthy elderly persons?

Participants will:

* Be characterized by means of: 1) evaluation of body composition, using anthropometric techniques, bioimpedance and 2) biochemical analyses: biochemical profile, lipid profile, serum ferritin, fasting glycemia, HbA1c and insulin.
* Arrive at fast to the laboratory and eat randomly control bread, 30% Chilean beans supplemented bread or glucose. Venous blood samples will be taken from the cubital fossa of the dominant arm at: 0, 30, 60 and 120 min postprandial, only after intake of bread control and supplemented bread. In addition, capillary blood will be taken at 0, 15, 30, 60, 90 and 120 min postprandial after intake of glucose, bread control or supplemented bread.

DETAILED DESCRIPTION:
Screening and initial characterization:

Initial screening: General health status will be consulted, and glycemia will be measured at any time, using a hemoglucotest. If eligible (glycemia at any time less than 140 mg/dL), the subjects will be invited to participate in the initial characterization and postprandial study.

Initial characterization:

A medical and nutritional evaluation will be carried out. A medical doctor will ask the volunteers for general information about their state of health and medication consumption.

The nutritional evaluation (weight, height, waist circumference and body composition) will be carried out in the Nutritional Status Evaluation Laboratory of the School of Nutrition and Dietetics of the University of Talca.

For the bioimpedance studies, volunteers will be asked prior to the assessment to:

* Do not drink alcohol 48 hours before the analysis.
* Having urinated 30 minutes before the analysis.
* Attend the laboratory on fasting, special care must be taken not to drink coffee 4 hours before the measurement.
* When the volunteers arrive at the laboratory, they will be asked to sit on a platform barefoot and without jewelry or metals, with the least amount of clothing possible (light clothing, light overalls, and a T-shirt to have a more exact weight, they will be asked to avoid wearing jeans that day).
* For the measurement of the waist circumference, the volunteers will be asked to lift their shirt or blouse, until their ribs or equivalent height can be seen. These measurements will be performed by a Nutritionist in an office to protect the privacy of the volunteers.
* Clinical laboratory blood samples. Participants will be informed by telephone of the day on which blood samples will be taken, for which they will be asked to eat their last meal at 11:00 p.m. the night before the blood test. The van will pick them up at their home, 11-12 people in total. The blood sample will be taken at the Fleming Clinic.
* Once the results are known, at least one week in advance, we will contact the volunteers by phone to make an appointment with the doctor and eat the first of four meals.

Food intake and blood sampling.

On the day of meal intake, volunteers will be asked to have their last meal at 11:00 p.m. the day before it will be presented in the laboratory. A van will pick up the volunteers between 6:30-8:00 a.m. They will be transferred to the Fleming Clinic along with 11-12 other people to the laboratory. Once in the laboratory, two types of blood samples will be taken:

1. Capillary blood: pricking a fingertip with a sterile lancet. A nutritionist will clean the finger of the volunteers with alcohol and later they will feel a slight prick, lasting less than a second. Capillary glycemia will be measured with that blood. This procedure will be carried out at times 0, 15, 30, 45, 60, 90 and 120 min after eating bread or glucose.
2. Venous blood: upon arrival at the laboratory (fasting) a Nurse will insert a conventional venous line in the arm. A 5 mL sample (equivalent to a teaspoon) of blood will be drawn at the following times: 0, 30, 60, and 120 min. Per day each volunteer will donate aprox. 20mL of blood, equivalent to approximately two tablespoons.

After arriving at the laboratory and taking the samples fasting (time 0), the volunteers will randomly receive one of the 2 samples of bread or glucose. If they receive glucose, only capillary blood samples will be taken.

If they receive a sample of bread, the volunteer must eat approximately 100 g (amount containing 50g of carbohydrates), (equivalent to 1 common bread) of the bread manufactured by us, along with 250 mL of water. Food intake time will be timed, and the volunteers should eat slowly but steadily. The intake time from the first bite to the last cannot exceed 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Persons between 60-70 years old.
* Persons autonomous.
* Persons who are willing to participate in this study and who have agreed and signed the informed consent.

Exclusion Criteria:

* Clinical diagnosis of diabetes
* Persons with levels of glycosylated hemoglobin (HbA1c) lhigher than 6.5
* Clinical diagnosis and uncontrolled chronic diseases.
* Anemia, dtermined by ferritin levels less than 15 µg/ L.
* Oropharyngeal disorders (self-reported).
* Persons with gastric bypass surgery.
* Celiac disease (self-reported).
* Coagulation disorders (self-reported).
* Use of medications that modify the glycemic response or lipid profile (acarbose, thiazolinediones, metformin, insulin, orlistat, among others).
* Clinical diagnosis of Alzheimer's disease or sinile dementia.
* People with pacemakers or metal subcutaneous implants.

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in the postprandial levels of methylglyoxal in plasma | 0, 30, 60 and 120 min postprandial
  Determiantion of the change in the levels of methylglyoxal in plasma by means of pre-column derivatization and posterior separation, detection and quantification by means of high performance liquid chromatography and detection by fluorescence

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Ávila, PhD, Principal Investigator — School of Nutrition and Dietetics, Health Sciences Faculty, University of Talca
Locations (1):
- School of Nutrition and Dietetics, Talca, Chile

IPD SHARING:
Plan to Share IPD: No
This was not authorized by the Institutional Ethics Comitee